CLINICAL TRIAL: NCT05952466
Title: Optical Coherence Tomography Angiography Evaluation of Retinal and Choroidal Microvascular Parameters in School-age Children in a COVID-19 Infection Pandemic Peak in China
Brief Title: Retinal and Choroidal Microvascular Parameters in School-age Children in a COVID-19 Infection Pandemic Peak in China
Status: Completed | Type: Observational
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Yuehong Zhang, Dr., Guangzhou First People's Hospital
Other Study IDs: GuangzhouFPH1
Record Dates: First submitted 2023-07-18; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19 infection; retinal microvascular involvement; choroidal thickness; school-age children
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 infection group: School-age children infected recently with COVID-19
- control group: School-age children without COVID-19

SUMMARY:
We designed this study to examine whether COVID-19 infection could lead to retinal and choroidal microvascular involvement in school-age children (6-18 years) in a pandemic peak in China.

DETAILED DESCRIPTION:
This is an observational case-control study. One hundred school-age children who visited the Department of Ophthalmology at Guangzhou First People's Hospital in China from February 1, 2023 to March 31, 2023 were included in this study. Eighty children with COVID-19 infection were included in the case group. Controls without COVID-19 infection were matched to COVID-19 infection cases by a ratio of 1:4 using frequency matching on age and gender. The primary end point of this study is the retinal and choroidal microvascular changes in school-age children during the COVID-19 pandemic. Secondary endpoint is the

ELIGIBILITY:
Inclusion Criteria:

Totally 100 school-age children (6-18 years) were enrolled in this study. All subjects had visited the ophthalmology clinic for routine ocular examinations. Refraction after ciliary muscle paralysis, myopia ≥ -6.0 spherical diopter, astigmatism ≤ 2.5 cylindrical diopter.

Exclusion Criteria:

1. The child or guardian did not agree to participate in the study.
2. Children could cooperate to complete the ocular examination.
3. The child had previous diseases affecting visual function and fundus, except for the diagnosis of refractive error.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Totally 100 school-age children (6-18 years) were enrolled in this study. All subjects had visited the ophthalmology clinic for routine ocular examinations.Eighty children with COVID-19 infection were included in the case group. Controls without COVID-19 infection were matched to COVID-19 infection cases by a ratio of 1:4 using frequency matching on age and gender. The following age subgroups were used for matching: 6-10, 10-14 and 15-18 years. A list of numbers computer-generated by a research member (Xu Zhang) was used to match the controls. The collected data included demographic and clinical data, as well as retinal and choroidal microvascular parameters.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Macular and peripapillary blood perfusion density | 5 minutes
  The blood flow density represents the proportion of the blood flow signal area in the scanning area to the overall area, expressed in units of mm-1, which can show the blood vessel perfusion and circulation.
Macular and peripapillary retinal thickness | 3 minutes
  Macular fovea and peripheral retinal thickness, retinal thickness around the optic nerve

SECONDARY OUTCOMES:
Fundus lesions | 2 minutes
  Such as fundus hemorrhage, exudation, vascular tortuous expansion, etc.
Vascular distribution shape in macular area | 2 minutes
  The measurement parameters of the foveal avascular zone include area, perimeter and non-circular index

CONTACTS AND LOCATIONS:
Overall Officials: Yuehong Zhang, Principal Investigator — Guangzhou First People's Hospital, Guangzhou, Guangdong China
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided